CLINICAL TRIAL: NCT02393482
Title: Psychological Impact of Amenorrhea in Women With Endometriosis: Perspective Randomized Study
Brief Title: Psychological Impact of Amenorrhea in Women With Endometriosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, MD,PhD, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMENORREA
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Amenorrhea; Endometriosis; Quality of Life
MeSH Terms: conditions — Amenorrhea; Endometriosis | interventions — Gonadotropin-Releasing Hormone; Leuprolide; tibolone; Calcium Carbonate; Cholecalciferol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balanced estroprogestins (Active Comparator): Women assigned to this arm will assume balanced monophasic estroprogestins (etinil-estradiol 100 mcg/levonorgestrel 20 mcg), one tablet orally daily, for 180 days.
  Interventions: Drug: Estroprogestinic therapy (Etinil-estradiol/levonorgestre)
- GnRHa (Active Comparator): Women assigned to this arm will assume Leuprorelin acetate (3,75 mg/2ml), one intramuscular administration every 28 days. After 45 days of treatment, therapy will be implemented with Tibolone 5 mg, one tablet daily orally, and Calcium carbonate/colecalciferol (500 mg/400 UI), one tablet daily orally. This therapy will be prosecuted for the remaining 135 days of treatment.
  Interventions: Drug: Gonadotropin-releasing hormone agonist (Leuprorelin acetate); Drug: Add back therapy 1 (tibolone); Drug: Add back therapy 2 (calcium carbonate/colecalciferol)

INTERVENTIONS:
Drug: Estroprogestinic therapy (Etinil-estradiol/levonorgestre) — Etinil-estradiol/levonorgestrel (100 mcg/20 mcg)/die
  Arms: Balanced estroprogestins
Drug: Gonadotropin-releasing hormone agonist (Leuprorelin acetate) — Leuprorelin acetate (3,75 mg/2 ml)/month
  Arms: GnRHa
Drug: Add back therapy 1 (tibolone) — tibolone 5 mg/die
  Arms: GnRHa
Drug: Add back therapy 2 (calcium carbonate/colecalciferol) — calcium carbonate/colecalciferol (500mg/400UI)/die
  Arms: GnRHa

SUMMARY:
The purpose of the study is to evaluate the impact on quality of life, psychological health, sexuality and chronic pain of therapies which determine amenorrhea in symptomatic women with endometriosis, through the administration of self reported questionnaires. Amenorrhea in the first group is caused by balanced assumption of estroprogestins, in the second group is caused by GnRHa-induced hypoestrogenism.

ELIGIBILITY:
Inclusion Criteria:

* Clinical, echographical or surgical diagnosis of endometriosis

Exclusion Criteria:

* Comorbidity
* Psychiatric diseases
* Refusal or inability to sign informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life (self reported questionnaires) | 180 days
  This outcome will be evaluated through self reported questionnaires
Sexual health (self reported questionnaires) | 180 days
  This outcome will be evaluated through self reported questionnaires
Psychological impact (self reported questionnaires) | 180 days
  This outcome will be evaluated through self reported questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari,Obstetrics and Gynecological Department,, Monserrato, Cagliari, Italy

REFERENCES:
- [Background] McWilliams LA, Cox BJ, Enns MW. Mood and anxiety disorders associated with chronic pain: an examination in a nationally representative sample. Pain. 2003 Nov;106(1-2):127-33. doi: 10.1016/s0304-3959(03)00301-4. PMID 14581119